CLINICAL TRIAL: NCT06128343
Title: Anatomical-Clinical Base of Adenocarcinoma Pancreatic
Acronym: BACAP-2
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/21/0191; 2021-A01050-41 (Other: ID-RCB)
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Adenocarcinoma; Carcinoma; Neoplasms
Keywords: Adenocarcinoma; fine-needle aspiration; endoscopic ultrasonography; epidemiology; biobank; DNA tumors
MeSH Terms: conditions — Adenocarcinoma; Carcinoma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample and micro-biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: collection of biological samples — Collection of biological samples including whole blood and micro-biopsy from tissue of pancreas

SUMMARY:
BACAP-2 is a prospective biobank dedicated to the pancreatic adenocarcinoma including clinical data and biological samples from tumor. The aim is to enrich the previous propective collection BACAP in order to support future research projects.

DETAILED DESCRIPTION:
Pancreatic cancer represents the fourth cause of death by cancer in Western countries. In over 90% of cases, it is due to an adenocarcinoma. The only curative treatment for pancreatic cancer remains the surgical exeresis. This one can only be suggested as a curative treatment in only 10 to 15% of cases. Besides, prevention or screening is difficult to set up due to the absence of clearly identified risk factors or groups and to the absence of useful markers for the diagnosis in clinical practice.

The research efforts in this area must face a double challenge: saving time while improving the diagnosis period and strengthen the therapeutic equipment. It is important to identify and characterise the new molecular markers applicable for a better diagnosis and/or treatment (especially the response factors to chemotherapy).

The present project aims to enrich with fresh tumor tissue and somatic genetic analysis the existing propective collection BACAP in order to support support future research projects on:

* the development of new diagnostic tools,
* understanding the development of tumors of the pancreas
* the development of new therapeutic targets
* understanding the response to chemotherapy…

ELIGIBILITY:
Inclusion Criteria:

* Patient with pancreatic mass syndrome explored by ultrasound endoscopy with cytopuncture or
* Patient with pancreatic mass syndrome explored by an abdominal scanner with and without injection of product contrast and/or puncture of the mass or secondary lesions by radiological route or
* Patient with pancreatic adenocarcinoma proven histologically and/or cytologically

Exclusion Criteria:

* Patient with a pancreatic tumor whose analysis histological is not an adenocarcinoma
* Pregnant or breastfeeding patient

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a pancreatic adenocarcinoma proven cytologically or histologically without any treatment
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2035-01-31 (Estimated); Study Completion 2035-02-28 (Estimated)

PRIMARY OUTCOMES:
Enrichment of prospective BACAP collection | 5 years
  This collection is coming to enrich the prospective BACAP collection of fresh tumor tissue and/or fixed from the micro-biopsy under endoscopic ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Barbara BOURNET, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (8):
- France (8):
  - Béthune hospital center, Béthune
  - Haut-Lévêque Hospital, Bordeaux
  - Huriez Hospital, Lille
  - Jean Mermoz private hosptila, Lyon
  - Saint Eloi Hospital, Montpellier
  - Regional Cancer Center From Montpellier, Montpellier
  - PAU hospital, Pau
  - Rangueil hospital, Toulouse

REFERENCES:
- [Derived] Bardol T, Dujon AM, Taly V, Dunyach-Remy C, Lavigne JP, Costa-Silva B, Kurma K, Eslami-S Z, Cayrefourcq L, Canivet C, Muscari F, Bournet B, Alix-Panabieres C. Early detection of pancreatic cancer by liquid biopsy "PANLIPSY": a french nation-wide study project. BMC Cancer. 2024 Jun 10;24(1):709. doi: 10.1186/s12885-024-12463-8. PMID 38853244